CLINICAL TRIAL: NCT06757166
Title: Effects of Early vs. Delayed Invasive Mechanical Ventilation: A Target Trial Emulation
Brief Title: The Effect of NOn-invasive Respiratory Support on outcoMe and Its Risks in SARS-COV-2-related Hypoxemic Respiratory Failure
Acronym: NORMO2
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Carmen Reep, PhD Candidate (MSc), Department of Intensive Care, Erasmus MC, Erasmus Medical Center
Other Study IDs: 50-56300-98-2113
Record Dates: First submitted 2024-12-23; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Target Trial Emulation, Invasive Mechanical Ventilation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endotracheal intubation — endotracheal intubation for invasive mechanical ventilation

SUMMARY:
To determine whether early endotracheal intubation compared to late endotracheal intubation affects clinical outcome (duration of invasive mechanical ventilation, mortality).

DETAILED DESCRIPTION:
Non-invasive respiratory support, especially HFNO is usually well-tolerated, especially in COVID-19 patients and can be applied for a prolonged period of time. However, there is a heated debate whether later/delayed endotracheal intubation (due to HFNO / NIV) increases the risk of lung injury, so-called patient self-inflicted lung-injury (P-SILI). The concept of P-SILI assumes that high forces applied to the lung resulting from strenuous breathing effort generated by the patient exacerbates lung-injury and is associated with adverse clinical outcome. It is therefore important to investigate if a longer period of non-invasive respiratory support before invasive mechanical ventilation is associated with adverse clinical outcome. Thus, it is unknown if delaying invasive ventilation worsens clinical outcome. In this study, the research question is whether early compared to late endotracheal intubation improves clinical outcome (duration of invasive mechanical ventilation, mortality)? The aim is to identify the optimal S/F ratio and respiratory rate thresholds for initiating intubation to either improve survival or reduce the duration of invasive ventilation without compromising survival. This is achieved by comparing 25 dynamic treatment regimes defined by combinations of S/F thresholds (<any, 250, 200, 150, 100) and respiratory rate thresholds (>any, 16, 20, 25, 30). Thresholds indicating less severe illness (e.g., S/F < 250 and RR > 16) are considered 'early intubation,' while thresholds indicating more severe illness (e.g., S/F < 100 and RR > 30) are considered 'late intubation'.

Two sensitivity analyses will be conducted:

1. Restricting to patients without hypercapnia (pCO2 < 45), excluding those with missing pCO2 values or pCO2 > 45.
2. Including only patients with non-missing Glasgow Coma Scale (GCS) values and adjusting for GCS as a confounder.

Additionally, seven subgroup analyses will be conducted:

1. Patients diagnosed with COVID-19
2. Patients with a history of COPD
3. Patients with a history of CHF
4. Patients with BMI ≤ 30
5. Patients with BMI > 30
6. Patients on high-flow nasal oxygen (HFNO) at time zero
7. Patients on non-invasive ventilation (NIV) at time zero

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized (inpatient or ICU)
* 18 years or older
* Hypoxemic respiratory failure: S/F<250
* Not yet intubated

Exclusion Criteria:

* Do not intubate order
* Presence of tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the United Stated for which data is registered in the National Covid Cohort Collaborative (N3C).
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
28-day RMTL of mortality | 28 days
  Mortality restricted mean time lost (RMTL) over the 28-day period (area under the cumulative incidence function curve)
28-day mortality risk | 28 days
  Mortality risk at day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Centre, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No